CLINICAL TRIAL: NCT04357665
Title: Laparoscopic Versus Open Mesh Repair of Bilateral Primary Inguinal Hernia 3 Armed Randomized Trial
Brief Title: Laparoscopic Versus Open Repair of Bilateral Primary Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohamed El Messiry, Ass. Professor of Surgery, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0302765
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Bilateral Inguinal Hernia; Postoperative Complications
Keywords: Bilateral Inguinal Hernia; Laparoscopic versus open mesh repair; Operative outcomes; Recurrence
MeSH Terms: conditions — Postoperative Complications; Recurrence

STUDY DESIGN:
Intervention Model Description: This prospective study included 120 consecutive patients with bilateral primary inguinal hernia managed by simultaneous bilateral repair. Patients were randomized by sealed opaque envelopes containing computer generated random numbers into 3 groups, each includes 40 patients. Group I treated by laparoscopic transabdominal preperitoneal repair using 2 separate meshes (Lap TAPP), Group II treated by open preperitoneal mesh repair with mesh fixation (Open PP), while Group III treated by standard bilateral Lichtenstein repair (LICHT group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lap TAPP Group (Active Comparator): Patients treated by laparoscopic transabdominal preperitoneal repair using 2 separate meshes fixed by laparoscopic tackers
  Interventions: Procedure: Bilateral TAPP Repair
- Open PP Group (Active Comparator): Patients treated by open preperitoneal single mesh repair fixated using sutures
  Interventions: Procedure: Open PP Repair
- Bilateral LICHT Group (Active Comparator): Patients treated by standard bilateral Lichtenstein repair using 2 separate meshes fixed by sutures
  Interventions: Procedure: Bilateral Lichtenstein Repair

INTERVENTIONS:
Procedure: Bilateral TAPP Repair — laparoscopic transabdominal preperitoneal repair using 2 separate meshes fixed by laparoscopic tackers
  Arms: Lap TAPP Group
Procedure: Open PP Repair — Open pre-peritoneal repair using single mesh fixed by sutures
  Arms: Open PP Group
Procedure: Bilateral Lichtenstein Repair — Bilateral Lichtenstein Repair using 2 separate meshes fixed by sutures
  Arms: Bilateral LICHT Group

SUMMARY:
Currently, there is a controversy regarding the best approach for simultaneous repair of bilateral inguinal hernia. The aim of this study was to compare the outcome of laparoscopic versus open repair of bilateral inguinal hernia

DETAILED DESCRIPTION:
This prospective randomized study included 120 consecutive patients with bilateral primary inguinal hernia treated at Alexandria university hospital in the period between June 2014 and February 2017. Patients were randomized by sealed envelopes into 3 groups, each includes 40 patients. Group I treated by laparoscopic transabdominal preperitoneal repair using 2 separate meshes, Group II treated by open preperitoneal mesh repair, while Group III treated by bilateral Lichtenstein repair. The 3 groups were compared regarding: operative time, postoperative complications, pain, hospital stay, return to normal activity and work, chronic groin pain, patient's satisfaction and 3 years recurrence rate.

Statistical Analysis: Numerical data in both groups was expressed as mean

± standard deviation (SD) and compared using One-way analysis of variance while categorical data was expressed as percentages and compared using Chi-squared test. Logistic regression test was used to determine predictors of postoperative complications. Differences were considered significant at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary bilateral inguinal hernias in patients aged from 20 to 60 years

Exclusion Criteria:

1. - Immune compromised patients,
2. - Morbid obesity (BMI > 35 kg/m2)
3. - Chronic liver or renal disease
4. - Coagulopathy
5. - High-risk patients unfit for major surgery (ASA III or IV)
6. - Recurrent hernias
7. - Complicated hernias
8. - Massive scrotal hernias
9. - Previous infra-umbilical surgery
10. Persistent groin pain due to other causes

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Operative time | Same day of surgery
  Operative time (in minutes)
Postoperative pain 7 days after surgery | 7 days after surgery
  Pain intensity was assessed using the pain visual analogue scale (VAS) with values ranging from 1 (no pain) to 10 (worst possible pain)
Early postoperative complications | 30 days after the surgery
  Any complications related to surgery developed within 30 days after the surgery

SECONDARY OUTCOMES:
Chronic postoperative pain | 3 months after surgery
  Groin pain related to surgery lasting for more than 3 months after surgery
Hernia recurrence | 3 years after surgery
  Unilateral or bilateral - residual or recurrent hernia within 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elmessiry, Principal Investigator — Ass. Professor of Surgery; Ahmed Gebaly, Principal Investigator — Ass. Professor of Surgery

IPD SHARING:
Plan to Share IPD: No
No consent to share IPD

REFERENCES:
- [Background] Feliu X, Claveria R, Besora P, Camps J, Fernandez-Sallent E, Vinas X, Abad JM. Bilateral inguinal hernia repair: laparoscopic or open approach? Hernia. 2011 Feb;15(1):15-8. doi: 10.1007/s10029-010-0736-2. Epub 2010 Oct 21. PMID 20960019
- [Background] Sarli L, Iusco DR, Sansebastiano G, Costi R. Simultaneous repair of bilateral inguinal hernias: a prospective, randomized study of open, tension-free versus laparoscopic approach. Surg Laparosc Endosc Percutan Tech. 2001 Aug;11(4):262-7. doi: 10.1097/00129689-200108000-00007. PMID 11525372
- [Background] Mahon D, Decadt B, Rhodes M. Prospective randomized trial of laparoscopic (transabdominal preperitoneal) vs open (mesh) repair for bilateral and recurrent inguinal hernia. Surg Endosc. 2003 Sep;17(9):1386-90. doi: 10.1007/s00464-002-9223-x. Epub 2003 Jun 17. PMID 12802653